CLINICAL TRIAL: NCT01058590
Title: Inflammatory Markers in Infants With Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Aviv Goldbart MD, Soroka UMC
Other Study IDs: SOR494810ctil
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Inflammation; Adenotonsillectomy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and urine will be obtained before therapy (T%A) snd 3 months afterwards. The serum will be stored at -70 throughout the study in the PI's Lab (DR.Goldbart) At the end of the study the sampled will be assessed for the presence of inflammatory markers (cytokines).

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is a common disorder in children (2-3%). OSAS in turn, is associated with significant behavioral, learning, and heart problems. Adenotonsillectomy (T&A, meaning the removal of tonsils and adenoids) is the most common treatment for the problem .Diagnosis of OSAS in children is based on overnight polysomnography (sleep study). Recent studies suggest that upper airway and systemic inflammatory changes exists in school-age children and adults with OSAS, and that anti inflammatory therapy can improve respiratory parameters during sleep and reduce adenoid size, similar to surgery. However, there are no data in the literature on inflammatory changes in infants with the disorder.

Healthcare resources utilization, a sensitive marker for diseases is consumed by young children (<3y) with OSAS more then healthy children, from their first year of life We hypothesize that infants and young children with OSAS present local inflammatory changes of the airways as well as systemic inflammation (in the blood or urine) that contribute to the learning, growing and heart associated medical problems. The Aims of the present study are to characterize the local and systemic inflammatory changes of young children with OSAS, and to evaluate their associated medical problems at diagnosis and after therapy (T&A) If indeed inflammation is "responsible" for the development of OSAS at such a young age it should be reduced following therapy (i.e. T&A). In such a case bio-markers may become a part of the algorithms for diagnosis and follow up of such patients.

DETAILED DESCRIPTION:
Specific Aims:

1. To conduct a trial evaluating the effect of Adenonsillectomy in infants (1-36 months of age), with OSA. Outcome measures will include polysomnographic findings conducted prior to and 12 weeks following surgery.
2. To identify the presence of inflammatory markers (such as, but not only Leukotriene B4, Leukotriene C4/D4/E4, Isoprostane-8, IL-6, TNF-alpha, and other pro inflammatory cytokines) in the peripheral blood (prior and after therapy), and urine (Leukotriene E-4, and others) and correlate their local and systemic expression prior and after therapy to the magnitude of therapy-associated response.

Study Duration: Two years (initial recruitment will be completed within the initial 12 months of the study). Assessment of the samples obtained throughout the study will be done at the latter part of the study.

Setting: Soroka University Hospital . The Sleep Laboratory in Soroka UMC, is the only pediatric one in the city of Beer Sheva and surroundings, evaluates over 1,000 children/year for a variety of sleep disorders, among which >700 are referred for suspected OSAS, among them 100 infants< 2 years/ year.

All children referred for surgery are admitted in the Dept. of Pediatrics where the PI works. We intend to approach all the children prior to surgery and offer them to participate in this study. Those who are interested will gain a sleep study following surgery to validate (or to rull out) the presence of residual OSA and if there is a need, to continue follow up in the pediatric sleep outpatient clinic in Soroka UMC.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month-3 years
* Diagnosis of obstructive sleep apnea syndrome(according to a sleep study)

Exclusion Criteria:

* Congenital disorders of the respiratory system
* Congenital craniofacial disorders (retrognathia, Trisomy 21)
* Use of anti inflammatory medications (like: montelukast, budesonide) up to 4 weeks prior to study entry.

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 0-3 years diagnosed with obstructive sleep apnea syndrome, refferred to removal of tonsills and adenoids
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Analysis of average change in inflammatory markers, before -to-after T%A. | February 2011

CONTACTS AND LOCATIONS:
Overall Officials: Aviv D Goldbart, MD, Principal Investigator — Soroka UMC
Locations (1):
- Soroka UMC, Beersheba, Israel

REFERENCES:
- [Background] Goldbart AD, Tal A. Inflammation and sleep disordered breathing in children: a state-of-the-art review. Pediatr Pulmonol. 2008 Dec;43(12):1151-60. doi: 10.1002/ppul.20943. PMID 19009600